CLINICAL TRIAL: NCT05140330
Title: French Tittle : Recherche Visant à améliorer l'ALimentation et l'Activité Physique du Sujet AGE Vivant à Domicile - Etude ALAPAGE
Brief Title: Improving Nutrition and Physical Activity in the Elderly Living at Home - ALAPAGE Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Observatoire Regional de la Sante Provence-Alpes-Côte d'Azur (Other)
Collaborators: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other); University of Avignon (Other); University of Bordeaux (Other); Caisse d'assurance retraite et santé au travail du Sud-Est (Unknown); Mutualité Française Sud (Unknown); Association santé éducation et prévention sur les territoires de Paca (Unknown); Institut de Recherche en Santé Publique, France (Other); Agence Régionale de Santé Provence-Alpes-Côte d'Azur (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-A03151-38
Record Dates: First submitted 2021-11-04; First posted 2021-12-01 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Nutrition, Healthy
Keywords: Elderly; Dietary diversity; Lifestyle integrated Functional Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 7 ALAPAGE sessions over 2 months and 1 evaluation session at 3 months
  Interventions: Behavioral: ALAPAGE workshop
- Control (Other): 3 evaluation sessions over 2 months and 1 session at 3 months
  Interventions: Behavioral: control workshop

INTERVENTIONS:
Behavioral: ALAPAGE workshop — 7 weekly group sessions over 2 months (1 introduction session, 2 physical activity sessions and 4 nutrition sessions) and 1 evaluation session at 3 months
  Arms: Intervention
Behavioral: control workshop — 3 evaluation group sessions over 2 months and 1 session at 3 months. After those 4 sessions, the participants will benefit from an ALAPAGE workshop
  Arms: Control

SUMMARY:
CONTEXT Promoting healthy aging and preventing loss of autonomy are critical issues for many countries. In France, the 2018-2022 national health strategy emphasizes that adequate nutrition and regular physical activity are key elements of healthy aging. Numerous prevention interventions to improve diet and physical activity in older adults exist in France and abroad, but very few have been evaluated. The ALAPAGE1 prefiguration study revealed a large number of preventive nutrition activities for seniors in Southeastern France, mainly as group prevention workshops. This study showed the need to i) improve the participation of socially isolated and/or economically vulnerable seniors in these workshops to avoid increasing social inequalities in health; ii) improve the form and content of the workshops and harmonize practices; and iii) evaluate the impact of these workshops. A strong partnership dynamic between our research teams and key players in the field of nutrition prevention for seniors has been initiated. It has enabled the co-construction of ALAPAGE project.

OBJECTIVES The main objective is to assess the impact of an improved prevention offer, the ALAPAGE group workshops, on the eating behaviors and physical activity of seniors living at home.

The secondary objectives are as follows:

* To assess the impact of seniors participation in the workshop on their feelings of loneliness and on their quality of life;
* To assess the mechanisms by which participation in a group workshop on diet and physical activity improves dietary diversity, physical ability and quality of life of participants, the acceptability of this workshop, the levers they activate and the psychosocial determinants of behaviour (intention, attitude, subjective norms, perceived control).

METHODS ALAPAGE workshops will be set up in local structures that usually receive elderly subjects for this type of activity. These workshops will be led by dieticians and professionals in adapted physical activity according to a protocol and with harmonized tools.

The intervention will take place according to the following phasing:

* Recruitment of the structures in which the 45 ALAPAGE workshops will take place
* Randomization of the workshops
* 30 Intervention workshops: 7 ALAPAGE sessions over 2 months and 1 evaluation session at 3 months
* 15 Control workshops: 3 evaluation sessions over 2 months and 1 session at 3 months
* Recruitment of 10 participants per workshop To answer the main objective, a dietary diversity score and the lower limb muscle strength will be assessed at the first session, the last session and 3 months after the last session, in both intervention and control participants. Others data will be collected throughout the workshop.

EXPECTED BENEFITS If the results of this research provide proof of concept that the prevention nutrition strategy based on ALAPAGE workshop, makes it possible, in the French context, to improve dietary diversity core and strength, this will constitute knowledge of major public utility. Participants will benefit from a personalized assessment of the diversity of their diet and their functional physical capacities and receive information and advice to adapt their diet and physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Be 60 years of age or older
* Live at home
* Understand French
* Be a beneficiary of a French social insurance scheme

Exclusion Criteria:

* Receive a personalized autonomy allowance.
* Have already participated in a preventive nutrition/physical activity workshop during the previous two years;
* Be under guardianship or curatorship.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Change in dietary diversity | First session, last session and 3 months after the last session, in both intervention and control participants
  Dietary diversity is assessed with the Diversity ALAPAGE Score (DAS). The DAS is calculated as follows: Consumption occurrences of 20 ALAPAGE food categories are reported from two 24H recall (for food eaten every day such as fruits, vegetables, meat excluding poultry, sweetened products, … ) and from a Food Frequency Questionnaire (FFQ, for foods which are consumed less often such as eggs, legumes, nuts, fatty fish, lean fish, and wholegrain cereals). According to the nutritional quality of its food category, each consumption earns negative or positive points. The DAS for one individual is the sum of all attributed points. A higher score means a greater dietary diversity. The DAS was recently applied to the dietary data of adults aged 60 years.old and over in a representative sample of the French population, and the distribution of the DAS was as follows: minimum = -40 ; mean = 53 ; maximum = 112 (Prat et al, 2021).
Change in lower limb muscle strength | First session and 3 months after the last session, in both intervention and control participants
  Assessed by a professional in adapted physical activity using the 30s chair-stand test (from the Senior Fitness Test)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Asept Paca, Marseille
  - Mutualité française Sud, Marseille

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prat,R., Gazan,R., Jacquemot, A.-F., Dubois, C., Feart,C., Darmon, N., Verger.E. Évaluation de la validité du score de diversité ALAPAGE avec des indicateurs de qualité nutritionnelle de l'alimentation de seniors en France (INCA3). Abstract JFN 2021
- [Derived] Bocquier A, Jacquemot AF, Dubois C, Trehard H, Cogordan C, Maradan G, Cortaredona S, Fressard L, Davin-Casalena B, Vinet A, Verger P, Darmon N; ALAPAGE Study Group; Arquier V, Briclot G, Chamla R, Cousson-Gelie F, Danthony S, Delrieu K, Dessirier J, Feart C, Fusinati C, Gazan R, Gibert M, Lamiraud V, Maillot M, Nadal D, Trotta C, Verger EO, Viriot V. Study protocol for a pragmatic cluster randomized controlled trial to improve dietary diversity and physical fitness among older people who live at home (the "ALAPAGE study"). BMC Geriatr. 2022 Aug 4;22(1):643. doi: 10.1186/s12877-022-03260-8. PMID 35927684